CLINICAL TRIAL: NCT01130389
Title: Trans-PBRN Case-control Study of Osteonecrosis of the Jaws
Brief Title: CONDOR Study of Osteonecrosis of the Jaws (TMJ)
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Gregg H. Gilbert, DDS, MBA, Study Chair, University of Alabama at Birmingham
Other Study IDs: 106037; U01DE016747 (NIH)
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Osteonecrosis of the Jaw
Keywords: ONJ

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to examine risk factors for osteonecrosis of the jaw (ONJ), including the possible association with bisphosphonates (BPs). This study used the research infrastructure from the three NIDCR-funded dental practice-based research networks (DPBRN, PEARL, PRECEDENT). De-identified data from the DPBRN were merged with comparable de-identified data from PEARL and PRECEDENT to form a single trans-PBRN data set used for analysis.

DETAILED DESCRIPTION:
The aims of this study were to (1) test the hypothesis that (BP) treatment is a risk factor for (ONJ); (2) to test the hypothesis that dental diseases (particularly periodontal disease), and invasive dental procedures such as dental extractions are true risk factors for (ONJ).

ELIGIBILITY:
Inclusion Criteria:

* participants directly involved in this study were patients of dentists from the dental practice based research networks (DPBRN, PEARL, PRECEDENT).

Exclusion Criteria:

* participants with a history of sickle cell anemia
* participants with a history of external severe trauma to the jaws

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The human subjects involved in this study were patients of dentists from the dental practice-based research networks (DPBRN, PEARL, PRECEDENT) who identified (ONJ) cases and chose to particpate in the study.
Sampling Method: Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H. Gilbert, DDS, MBA, Study Chair — Dental Practice-Based Research Network (DPBRN); Andrei Barasch, DMD, MDSc, Principal Investigator — Dental Practice-Based Research Network (DPBRN)
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon